CLINICAL TRIAL: NCT01270542
Title: Effect of Pre-operative Adjunctive Anti-VEGF on Growth Factors in Severe Proliferative Diabetic Retinopathy Requiring Surgical Management
Brief Title: Avastin for PDR (Proliferative Diabetic Retinopathy)
Acronym: PDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USC-HS-09-00068
Record Dates: First submitted 2010-12-01; First posted 2011-01-05 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2014-05

CONDITIONS: Retinal Detachment; Diabetic Retinopathy
Keywords: Traction Retinal Detachment (PDR); Proliferative Diabetic Retinopathy (PDR)
MeSH Terms: conditions — Retinal Detachment; Diabetic Retinopathy | interventions — Bevacizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avastin Injection Group (AIG) (Experimental): Subjects in this group will get single 0.05 mL intravitreal injection of bevacizumab 1.25 mg 3-7 days prior to surgery for tractional retinal detachment secondary to Proliferative Diabetic Retinopathy.
  Interventions: Drug: Avastin (bevacizumab)
- Sham Injection Group (SIG) (Sham Comparator): Subjects in this group will get a sham injection 3-7 days prior to surgery for tractional retinal detachment secondary to Proliferative Diabetic Retinopathy.
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Avastin (bevacizumab) — single 0.05 mL intravitreal injection of bevacizumab 1.25 mg
  Other Names: Avastin
  Arms: Avastin Injection Group (AIG)
Other: Sham injection — Subject's eyes will be anesthetized but no injection will be performed.
  Other Names: Sham
  Arms: Sham Injection Group (SIG)

SUMMARY:
The purpose of this study is to determine the effect of anti-VEGF drug (Avastin) adminstration in eyes prior to surgical treatment for Traction retinal detachment (TRD) in patients with Proliferative Diabetic Retinopathy (PDR).

DETAILED DESCRIPTION:
Traction retinal detachment (TRD) due to proliferative diabetic retinopathy is a blinding disease caused by contraction of fibrovascular proliferation, treatment of which is limited to surgery. Fibrosis and neovascularization are both associated with high levels of connective tissue growth factor (CTGF) and vascular endothelial growth factor (VEGF) in the eye. Small, nonrandomized studies have suggested that pre-operative adjunctive anti-VEGF administration may reduce intra- and post-operative complications and provide visual benefit in patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Active fibrovascular proliferation due to PDR with TRD given pre-operative clearance for pars plana vitrectomy (PPV) and TRD repair.

Exclusion Criteria:

* Dense vitreous hemorrhage
* Inability to follow-up for surgery within 3-7 days after intravitreal injection
* History of stroke, thromboembolic event, or heart attack within the last 6 months
* Less than 18 years of age
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Eliott, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074
- [Derived] Sohn EH, He S, Kim LA, Salehi-Had H, Javaheri M, Spee C, Dustin L, Hinton DR, Eliott D. Angiofibrotic response to vascular endothelial growth factor inhibition in diabetic retinal detachment: report no. 1. Arch Ophthalmol. 2012 Sep;130(9):1127-34. doi: 10.1001/archophthalmol.2012.1611. PMID 22965588

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Avastin Injection Group (AIG) | Sham Injection Group (SIG)
Started | 10; 10 Eyes | 9; 10 Eyes
Completed | 9; 9 Eyes | 8; 9 Eyes
Not Completed | 1; 1 Eyes | 1; 1 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Avastin Injection Group (AIG) | Sham Injection Group (SIG) | Total
Number analyzed (Participants) | 10 | 9 | 19
Number analyzed (Eyes) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 49 [31 to 62] | 53 [46 to 64] | 52 [31 to 64]
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 2 | 6 | 8
  Male | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Effect of an Anti-VEGF (Vascular Endothelial Growth Factor) Agent, Bevacizumab, on Levels of Vitreous and Aqueous Growth Factor Levels (pg/mL) in Eyes With Traction Retinal Detachment Due to PDR
Description: Comparison of vitreous VEGF levels (pg/mL) and aqueous VEGF (pg/mL) levels in bevacizumab and control groups.
Time Frame: 3 months after last surgery
Measure: Median (Full Range); unit: pg/mL
Units Other Than Participants: Eyes
Groups:
- Avastin (Bevacizumab): Subjects in this group will get single 0.05 mL intravitreal injection of bevacizumab 1.25 mg 3-7 days prior to surgery for tractional retinal detachment secondary to Proliferative Diabetic Retinopathy.
- Sham Injection: Subjects in this group will get a sham injection 3-7 days prior to surgery for tractional retinal detachment secondary to Proliferative Diabetic Retinopathy.
Arm/Group | Avastin (Bevacizumab) | Sham Injection
Number analyzed (Participants) | 10 | 9
Number analyzed (Eyes) | 10 | 10
pg/mL
  Vitreous VEGF levels | 0 [0 to 559] | 373 [0 to 1073]
  Aqueous VEGF levels | 13 [0 to 1652] | 0 [0 to 868]

2. Secondary Outcome: Whether Intra- and Post-operative Complications Are Decreased in Eyes Given Pre-operative Adjunctive Bevacizumab in Eyes Undergoing Proliferative Form of Diabetic Retinopathy (PDR) Surgery.
Time Frame: 3 months after last surgery.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Avastin (Bevacizumab) | Sham Injection
Number analyzed (Participants) | 10 | 9
Number analyzed (Eyes) | 10 | 10
Eyes
  Cataract | 1 | 1
  Vitreous hemorrhage | 0 | 1
  Ischemia | 0 | 2
  Glaucoma | 0 | 1

3. Secondary Outcome: Improvement of Visual Outcomes in Patients Given Pre-operative Adjunctive Bevacizumab in Eyes Undergoing PDR Surgery.
Description: Measured by median logMAR change in the best corrected visual acuity (VA) from baseline to post operative month 3 (POM3)
Time Frame: 3 months from last surgery
Measure: Median (Full Range); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Avastin (Bevacizumab) | Sham Injection
Number analyzed (Participants) | 10 | 9
Number analyzed (Eyes) | 10 | 10
logMAR | -0.18 [-2.0 to 1.0] | 0 [-1.0 to 4.4]

ADVERSE EVENTS:
Time Frame: 3 months after surgery
Arm/Group | Avastin Injection Group (AIG) | Sham Injection Group (SIG)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No